CLINICAL TRIAL: NCT04254276
Title: Musculoskeletal Pain of Neck and Shoulder Area in Female Office Workers: Relations Between Muscle Tone, Stiffness, Pain-pressure Threshold, Self-reported Pain Intensity and Physical Activity.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Martin Argus, MSc, University of Tartu
Other Study IDs: UTSP001
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Musculoskeletal Pain; Neck Pain; Shoulder Pain
Keywords: Musculoskeletal pain; Muscle tone; Muscle stiffness; Pain-pressure threshold; Neck; Shoulder; Office work
MeSH Terms: conditions — Musculoskeletal Pain; Neck Pain; Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic group: Office workers with neck and shoulder area musculoskeletal pain
- Asymptomatic group: Office workers without neck and shoulder area musculoskeletal pain

SUMMARY:
The objective of this study is to determine the differences between neck and shoulder region skeletal muscle tone, stifness, pain-pressure threshold, self-reported pain intensity and physical activity in female office workers. 50-100 participants aged 20-60 are anticipated.

DETAILED DESCRIPTION:
The objective of this study is to determine the differences between neck and shoulder region skeletal muscle tone, stifness, pain-pressure threshold, self-reported pain intensity and physical activity.

Participants: 50-100 subjects, all female, aged 20-60 are anticipated.

Methods: Skeletal muscle tone and stiffness are measured using myotonometry. Pain-pressure threshold is measured using algometry. Prevalence of neck and shoulder area musculoskeletal pain is recorded using Nordic questionnaire. Self-reported pain intensity is measured using VAS scale. Self-reported physical activity is recorded using Baecke physical activity questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Office work (at least 4 day per week, 8 hours a day with over 50% working with a computer)

Exclusion Criteria:

* Prior neck trauma, neurological or oncological conditions, recent use of muscle relaxants or painkillers, obesity (BMI of >30)

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50-100 subjects are anticipated, all female, aged 20-60. Office work of at least 4 days per week with over 50% of time working with a computer is required.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between muscle tone, stiffness and self-reported pain | March 1st 2020 - May 1st 2021
  Correlation between muscle tone (Hz), stiffness (N/m) of upper trapezius, levator scapulae and paraspinal upper neck muscles and self-reported neck and shoulder region pain intensity (VAS).

SECONDARY OUTCOMES:
Relationship between muscle tone, stiffness and pain-pressure threshold | March 1st 2020 - May 1st 2021
  Correlation between muscle tone (Hz), stiffness (N/m) and pain-pressure threshold (kPa) of upper trapezius, levator scapulae and paraspinal upper neck muscles in symptomatic and asymptomatic subjects.

IPD SHARING:
Plan to Share IPD: Undecided